CLINICAL TRIAL: NCT06720766
Title: Assessment of FibbroScan in Diagnosing MASLD Among the Chinese Population With Obesity
Acronym: MASLD
Status: Recruiting | Type: Observational
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hongmei Zhu, Assistant Researcher, The Third People's Hospital of Chengdu
Other Study IDs: 2023-S-177; CSY-YNXM-2023-001 (Other Grant/Funding Number: The Third People's Hospital of Chengdu)
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FibbroScan and biopsy — In individuals with obesity, a biopsy is performed within a week after undergoing an FibroScan examination.

SUMMARY:
The non-invasive evaluation of liver steatosis and fibrosis with FibroScan is a routinely procedure in clinical practice for people with obesity. However, there are still considerable uncertainties regarding the potential influence of confounding factors and the optimal application of cut-off values for obesity.

The goal of this observational study is to learn about the optimal application of cut-off values of for Chinese people with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older who provided written informed consent
2. Patients who schedule to undergo bariatric surgery and a liver biopsy (LB) for the investigation of suspected MASLD
3. Patients who schedule to undergo FibroScan examination

Exclusion Criteria:

1. Patients with ascites or pregnant women
2. Patients with any active implantable medical device (such as a pacemaker or defibrillator)
3. Patients who have undergone liver transplantation
4. Patients with cardiac failure and/or significant valvular disease
5. Patients with haemochromatosis
6. Patients who have refused to undergo LB or blood tests
7. Patients with a confirmed diagnosis of active malignancy, or other terminal disease
8. Patients participating in another clinical trial within the preceding 30 days

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients aged 18 years or older who provided written informed consent and were scheduled to undergo bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Through study completion, an average of 1 year
  Estimated using the area under the receiver operating characteristic curves for the categories of steatosis and fibrosis
Cut-off values | Through study completion, an average of 1 year
  Optimal thresholds for application on people with obesity

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Chengdu, Chengdu, Sichuan, China